CLINICAL TRIAL: NCT01984073
Title: Effect of Niacin On Fatty Acid Trapping
Brief Title: Effects of Niacin On Fatty Acid Trapping
Acronym: NOFAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Arizona Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Richard Dunbar, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NOFAT; K23HL091130 (NIH)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Dyslipidemia
Keywords: Atherogenic dyslipidemia phenotype
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ER Niacin Oral Fat Challenge (Active Comparator): ER Niacin (Niaspan) 2000mg one hour prior to Oral Fat Challenge using fresh cream at a dose of 50 g fat per square meter of body surface area. This is followed by frequent plasma and urine collections for next 12 hours to assess markers of fat metabolism and inflammation.
  Interventions: Drug: ER Niacin Oral Fat Challenge
- IR Niacin Oral Fat Challenge (Active Comparator): Immediate-Release Niacin (Nialor) 500 mg one hour prior to Oral Fat Challenge and again 1, 3 and 5 hours after the oral fat load for a total dose of 2 grams.Subjects will undergo plasma and urine collections for 12 hours to assess markers of fat metabolism and inflammation.
  Interventions: Drug: IR Niacin Oral Fat Challenge
- Placebo Oral Fat Challenge (Placebo Comparator): Placebo one hour before and 1,3, and 5 hours after oral fat load using heavy cream at 50 grams of fat per square meter of body surface area. Plasma and urine collections for 12 hours
  Interventions: Other: Placebo Oral Fat Challenge

INTERVENTIONS:
Drug: ER Niacin Oral Fat Challenge — Extended release niacin 2000 mg at hour 0, followed by oral fat challenge at hour 1.
  Other Names: Niaspan
  Arms: ER Niacin Oral Fat Challenge
Drug: IR Niacin Oral Fat Challenge — Nialor(R) 500mg or Placebo at hour 0, 2, 4, and 6. Oral fat challenge at hour 1 (one hour after first dose of immediate-release niacin)
  Other Names: Nialor
  Arms: IR Niacin Oral Fat Challenge
Other: Placebo Oral Fat Challenge — Placebo at hour 0. Oral fat challenge at hour 1, followed by placebo at hours 2,4,and 6
  Arms: Placebo Oral Fat Challenge

SUMMARY:
The purpose of this study is to understand whether a vitamin called NIcotinic ACid vitamIN (NIACIN for short, also known as vitamin B3) helps the body process dietary fat more efficiently. This is important because people with dyslipidemia have a problem with how they process fat, which raise the risk of heart disease.

DETAILED DESCRIPTION:
This study includes three phases, which each have a separate purpose. At this time, we are only recruiting for Phase 2. The purpose of this particular phase is to measure the effects of niacin after drinking a glass of heavy cream as a source of fat. We hope that studying the way the body responds will help us better understand how niacin works.

In this study, we are interested in niacin's ability to lower triglycerides, or fat in the blood. We are studying two different forms of niacin and comparing them to each other. The two forms differ in how long they take to release niacin into the bloodstream. The first form is called Nialor, and is sometimes called immediate-release niacin because it is absorbed into the bloodstream quickly. The second form is called Niaspan, and is sometimes called extended-release niacin because it is a time-released spansule that takes longer to get into the bloodstream. We are comparing the two forms because we think that the time that it takes to absorb niacin may affect how it works. We also want to understand one of the common effects of niacin: skin flushing. Most people who take niacin experience flushing, which is a hot flash. In this study, we are studying whether the two forms of niacin cause different degrees of flushing. Niaspan is approved by the US Food and Drug Administration (FDA) to treat unfavorable cholesterol levels and prevent heart attacks in those who have already suffered heart attacks. Nialor is available over the counter as a supplement and contains Silymarin (milk thistle) and Policosanol (an extract from sugar cane) in addition to niacin.

ELIGIBILITY:
Inclusion Criteria:

* Meet protocol defined criteria for atherogenic dyslipidemia phenotype
* Men and non-pregnant, non-lactating women between the ages of 22 and 75
* Fasting triglycerides <500 mg/dL
* Ability to understand and agree to informed consent
* Willingness to comply with study-related procedures

Exclusion Criteria:

* Dysbetalipoproteinemia
* History of extreme triglyceridemia (TG >500 mg/dL) or pancreatitis from triglyceridemia, regardless of whether it is currently controlled
* LDL >190 mg/dL
* History of chronic renal insufficiency (serum creatinine >2.0 mg/dL)
* History of non-skin malignancy within the previous 5 years
* Subject reported history of HIV
* Uncontrolled thyroid disease
* Hypoalbuminemia (serum albumin >2.5 mg/dL)
* Exposure to an investigational drug within 6 weeks prior to the screening visit
* Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition
* Major surgery within the previous 6 weeks
* Subjects who have undergone any organ transplant
* History of drug abuse within the past 3 years, or regular alcohol use >14 drinks per week
* Women who are breast-feeding
* Women who are pregnant by urine pregnancy test at each visit
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
* Change in statin dose within 6 weeks of the first experimental visit
* Use of the following non-statin lipid-altering therapy within 6 weeks of the first experimental visit: Niacin > 100 mg/day (Niacor, Slo-Niacin, Niaspan, Advicor, or supplemental niacin), Fibrates [gemfibrozil (Lopid), fenofibrate (Antara, Lofibra, Tricor, Triglide)], Enterically active drugs [colestipol (Colestid), cholestyramine (Questran), colesevelam (Welchol), ezetimibe (Zetia, Vytorin)], Red yeast rice, Fish oil (Omacor, numerous supplements)
* Use of medications indicated for the treatment of diabetes within 6 weeks of the screening visit
* Known intolerance or contraindication to niacin (e.g., moderate to severe gout, severe peptic ulcer disease)
* Medical condition that would prohibit fasting (e.g., diagnosis of insulinoma or postabsorptive hypoglycemia)
* Significant disinclination to dairy products (e.g., lactose intolerance, inviolable dietary restrictions)
* History of anaphylactic reaction
* For indocyanine green substudy: iodine allergy or shellfish allergy (n.b. a subject with an allergy can participate in the overall experiment, but will forego the indocyanine green tracer study)
* Donation of blood 8 weeks and/or treatment with medications for psychiatric disorders
* Hemoglobin <10 g/dL

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Plasma Triglycerides | Baseline to 12 hour post dose
  Plasma Triglycerides (TGs) after oral fat challenge will be measured to assess post-prandial lipidemia after niacin and placebo. Parameters of interest are the area under the curve (AUC), time to peak (t-max), and peak concentration (c-max). The relevant units will be mg.h/dl for plasma triglyceride AUC, minutes for time to peak plasma TG and mg/dl for c-max.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Dunbar, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Presbyterian Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No